IRB Protocol Number: 2022B0242 IRB Approval date: 8/2/2022

Version: 1

# The Ohio State University Consent to Participate in Research

**Study Title:** Strategies for Coping with Negative Thoughts

**Researcher:** Daniel R. Strunk, Ph.D.

**Sponsor:** None

3

1

- 4 This is a consent form for research participation. It contains important information about
- 5 this study and what to expect if you decide to participate.
- 6 Your participation is voluntary.
- 7 Please consider the information carefully. Feel free to ask questions before making your
- 8 decision whether or not to participate. If you decide to participate, you will be asked to sign
- 9 this form and will receive a copy of the form.

10 11

**Purpose:** The purpose of this study is to evaluate the effects of different approaches to coping with negative automatic thoughts.

12 13 14

15

16

17

18

**Procedures/Tasks:** First, we will ask you to complete a series of surveys asking about you and your day-to-day thoughts and feelings. Next, you will watch a few brief informational videos and then practice the strategies covered in the videos using a worksheet. You will then be contacted (by text or email) and sent one survey per day for 6 days, which will include a worksheet for you to complete. Approximately one week after completing the initial survey, you will be asked to complete another set of surveys.

19 20 21

**Duration:** Part one of this study will take about 60 minutes. The six daily surveys will take 5 minutes each for a total of 30 minutes. The final survey one week after starting the study will take 30 minutes. Thus, the total duration for your participation will be about 2 hours.

232425

26

27

22

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University.

28 29 30

31

**Risks and Benefits:** You will be asked questions about your mood and emotions, some of which may be uncomfortable for some people. You can skip any questions that you do not want to answer. There are no benefits to participation in the study.

323334

IRB Protocol Number: 2022B0242
IRB Approval date: 8/2/2022
Version: 1

#### **Confidentiality:**

35 36

> We will work to make sure that no one sees your survey responses without approval. But, because we are using the Internet, there is a chance that someone could access your online responses without permission. In some cases, this information could be used to identify you. Your data will be protected with a code to reduce the risk that other people can view the responses.

42 43

44

45

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law. Also, your records may be reviewed by the following groups (as applicable to the research):

46 47 48

• Office for Human Research Protections or other federal, state, or international regulatory agencies;

49 50 The Ohio State University Institutional Review Board or Office of Responsible Research Practices;
Authorized Ohio State University staff not involved in the study may be aware that

515253

you are participating in a research study and have access to your information; and

The sponsor, if any, or agency (including the Food and Drug Administration for FDAregulated research) supporting the study.

545556

**Future Research:** Your de-identified information may be used or shared with other researchers without your additional informed consent.

575859

60

61

62

63

64

**Incentives:** Participants can earn up to 2.0 REP credit hours. Credit will be awarded as follows: 1.0 credit for time 1, 0.5 credits for the daily surveys, and 0.5 credits for time 2. In order to earn each participation credit, you will need to respond correctly to attention checking items in the study. These should be straight forward to answer correctly as long as you are paying attention. Daily surveys should be completed by the end of the day (11:59pm) on which they are sent. Students can miss one daily survey and still obtain credit for the daily surveys.

656667

## **Participant Rights:**

68 69

70

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.

71 72 73

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

75 76 77

78

74

An Institutional Review Board responsible for human subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to

CONSENT
Behavioral/Social Science

IRB Protocol Number: 2022B0242 IRB Approval date: 8/2/2022

Version: 1

applicable state and federal regulations and University policies designed to protect the rights and welfare of research participants.

### **Contacts and Questions:**

81 82 83

For questions, concerns, or complaints about the study, or you feel you have been harmed as a result of study participation, you may contact Dr. Daniel Strunk at strunk.20@osu.edu.

848586

87

88

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact the Office of Responsible Research Practices at 1-800-678-6251.

89

## **Providing consent**

90 91 92

93

94

I have read (or someone has read to me) this page and I am aware that I am being asked to participate in a research study. I have had the opportunity to ask questions and have had them answered to my satisfaction. I voluntarily agree to participate in this study. I am not giving up any legal rights by agreeing to participate.

95 96 97

To print or save a copy of this page, select the print button on your web browser.

98 99

Please click the button below to proceed and participate in this study. If you do not wish to participate, please close out your browser window.

100 101